CLINICAL TRIAL: NCT04197882
Title: An Open-Label, Phase Ib Clinical Study to Evaluate OrienX010 in Combination With Toripalimab as Neoadjuvant Treatment in the Patients With Complete Resectable Stage III and Stage IV (M1a) Melanoma
Brief Title: Clinical Study to Evaluate OrienX010 in Combination With Toripalimab as Neoadjuvant Treatment in Advanced Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OrienX010-II-12
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
Keywords: complete resectable; melanoma; neoadjuvant treatment
MeSH Terms: conditions — Melanoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): This study consisted of 3 stage of neoadjuvant treatment, surgical, and adjuvant treatment. Neoadjuvant treatment period: OrienX010 intratumoral injection in combination with Toripalimab infusion. Toripalimab : 3 mg/kg, IV infusion: Once every 2 weeks for 6 doses ; OrienX010: Maximum injection volume 8 × 108 pfu, intratumoral injection: Once every 2 weeks for 6 doses ; Surgical treatment period: 2 weeks after the last dose of neoadjuvant treatment (± 7 days), the investigator designed the surgical protocol of the melanoma radical surgery according to the patient's individual disease, and performed postoperative care according to the patient's condition.
  Adjuvant treatment period: 3 weeks after operation (± 7 days), the patient was given Toripalimab infusion. Toripalimab 3 mg/kg intravenously given every 3 weeks (every 3 weeks per cycle) for up to 1 year (the one-year duration will be counted from 1st dose in neoadjuvant treatment).
  Interventions: Biological: OrienX010 Combination with Toripalimab injection

INTERVENTIONS:
Biological: OrienX010 Combination with Toripalimab injection — OrienX010 Produced by Oriengene Biotechnology Co.,Ltd. Strength: 1.0 mL/vial. Toripalimab infusion Produced by Junshi Biosciences Co., Ltd. Strength: 240 mg/6 mL/vial; Sterile water injection dosage form; Expiry date: 24 months; Date of manufacture: Based on the date of manufacture indicated in the product package.
  Other Names: Recombinant Human GM-CSF Herpes Simplex Virus intratumoral Injection combination with Recombinant Human Anti-PD-1 Monoclonal Antibody infusion

SUMMARY:
This study is an open-label, Phase Ib clinical study to evaluate recombinant human GM-CSF herpes simplex virus intratumoral injection (OrienX010) in combination with recombinant humanized anti-PD-1 monoclonal antibody infusion (Toripalimab) as neoadjuvant treatment in patients with complete resectable stage III and IV (M1a) melanoma.

This study is planned to enroll approximately 30 patients with stage III and IV melanoma (M1a) who meet protocol requirements.

This study is to evaluate the efficacy and safety of recombinant human GM-CSF herpes simplex virus intratumoral injection (OrienX010) in combination with recombinant humanized anti-PD-1 monoclonal antibody infusion (Toripalimab infusion) as neoadjuvant treatment in the patients with complete resectable stage III and IV (M1a) melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. An ICF approved by the Ethic Committee will voluntarily signed by the patient prior to initiating any screening or specific study procedures;
2. Male or female patients between 18 and 75 years of age;
3. Patients with definite diagnosis of complete resectable stage III and IV melanoma (M1a) based on histology and/or cytology, and with at least 1 measurable lesion(s).
4. Patients with ECOG performance status of 0 or 1;
5. Expected Survival> 4 months;

The patient has good function in each organ, and the following conditions are required at screening according to the laboratory reference range:

* White blood cell count ≥ 3.0 × 109/L;
* Absolute neutrophil value ≥ 1.5 × 109/L;
* Platelet count ≥ 100 × 109/L;
* Hemoglobin ≥ 90 g/L;
* Serum albumin ≥ 2.5 g/dL;
* Liver function tests: Total bilirubin ≤ 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN;
* Renal function tests: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min at 24 hours (Cockcroft and Gault formula);
* International normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (APTT) or partial prothrombin time (PTT) ≤ 1.5 × ULN;

  7. Female patients with childbearing potential (including premature menopause, menopausal < 2 years and non-surgical sterilization), male patients, and partners of male patients must agree to use effective contraception during the study: Surgical sterilization, oral contraceptives, intrauterine devices, sexual abstinence or barrier contraceptive combination spermicides; All patients must continue contraception for 6 months after the last treatment.

Exclusion Criteria:

1. Patients previously treated with T-VEC or similar; Patients previously treated with anti PD-1 antibody, anti PD-L1 antibody, anti PD-L2 antibody or similar;
2. Patients with negative anti-herpes simplex virus type I (HSV-1) antibodies IgG and IgM ;
3. The patient's lesion does not meet the requirement of the intratumoral injection volume or is not suitable for intratumoral injection;
4. Received anti-herpes simplex virus therapy (such as aciclovir, ganciclovir, valaciclovir, and arabinoside) within 4 weeks prior to the first dose of study treatment;
5. Received another anti-tumor monoclonal antibody (mAb) within 4 weeks prior to the first dose of study treatment or hasn't recover (≤ Grade 1) from adverse events due to prior therapy (occurring earlier than 4 weeks) ;
6. Patients with a history of other (including unknown primary) malignancies within 5 years prior to the first dose of trial treatment. Note: Except for fully treated stage 1 or 2 basal/squamous cell carcinoma of the skin, superficial bladder cancer, or in situ cancer that is treated with potentially curative therapy;
7. Patients with known hypersensitivity to the study drug, its active ingredient, excipients;
8. Patient with HBsAg positive and HBV DNA copies > 1×103copies/mL;
9. Patients with positive hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies;
10. Patients with any unstable systemic disease, including but not limited to: Serious infection, uncontrolled diabetes mellitus, unstable angina, cerebrovascular accident or transient cerebral ischemia, myocardial infarction, congestive heart failure, and serious arrhythmia liver, kidney, or metabolic disease requiring medical treatment;
11. patients with active CNS metastases. patients may participate in the study if their CNS is adequately treated and their neurological symptoms recover to levels less than or equal to Grade 1 (CTCAE) for at least 2 weeks before enrollment, with the exception of residual signs or symptoms associated with CNS therapy . In addition, patients must be those who do not use corticosteroids or who take stable doses of ≤ 10 mg prednisone/day (or equivalent dose) or who decrease to ≤ 10 mg prednisone/day;
12. Patients with autoimmune disease, received liver or other organs transplantation once before, active pulmonary tuberculosis; or patients received major surgical procedures, live vaccination, immunotherapy 4 weeks prior to study initiation
13. Tumor's macrovascular invasion in the iliac and femoral vessels;
14. The disease (e.g., mental illness, etc.) or condition (e.g., alcoholism or drug abuse, etc.) of the patient may increase the patient's risk of receiving trial medication or affect the patient's compliance with the study requirements, or may confuse the study results;
15. Within 30 days of screening, the patient had received any other study product or had participated in another intervention clinical trial;
16. Pregnant or lactating women, or women who are prepared to become pregnant or lactating during the study; Men or women who are unwilling to use effective contraception;
17. Other situations that the investigators think are not suitable for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-05-27 (Estimated); Study Completion 2025-05-27 (Estimated)

PRIMARY OUTCOMES:
pathological response rates | 12 week of treatment
  pCR and Major PR/Near pCR rates
Clinical effective rate | 12 week of treatment
  objective response rates based on RECIST 1.1, include CR,PR,SD

SECONDARY OUTCOMES:
RFS | 1-year and 2-year after surgery
  To evaluate 1-year relapse-free survival (RFS) and 2-year relapse-free survival
OS | approximate 3 years
  overall survival
the safety of OrienX010 in combination with Toripalimab | From date of enrolling to 90 days after end of treatment
  Number of participants with treatment-related SAE and adverse events that assessed by CTCAE v5.03
The surgical operation related events were observed | Surgical treatment period
  observe the surgical operation related events
Clinical effective rate | 12 week of treatment
  Objective response rates based on iRECIST and it-RECIST, include CR,PR,SD

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu J, Wang X, Li Z, Gao S, Mao L, Dai J, Li C, Cui C, Chi Z, Sheng X, Lai Y, Tan Z, Lian B, Tang B, Yan X, Li S, Zhou L, Wei X, Li J, Guo J, Si L. Neoadjuvant oncolytic virus orienx010 and toripalimab in resectable acral melanoma: a phase Ib trial. Signal Transduct Target Ther. 2024 Nov 22;9(1):318. doi: 10.1038/s41392-024-02029-2. PMID 39572525